CLINICAL TRIAL: NCT01392781
Title: Markers and Calculation of Cardiovascular Risk in the Distinct Phenotypes of Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Daskalopoulos Georgios, Aristotle University of Thessaloniki
Other Study IDs: 14/1-3-2011
Record Dates: First submitted 2011-07-06; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; hsC-RP; Lp-PLA2; cardiovascular risk
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- normoweight PCOS patients
- normoweight controls
- overweight plus obese PCOS patients
- overwqeight plus obese controls

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder and cause of anovulatory infertility among reproductive aged women. According to the revised criteria of 2003, four distinct phenotypes of PCOS can be diagnosed. However, there are emerging evidence supporting the existence of different levels of cardiometabolic risk between the four phenotypic groups of the syndrome. The purpose of this study is to determine the cardiovascular risk of i) normoweight and ii)overweight plus obese women of every one of the four phenotypes of the syndrome as well as the levels of low inflammation serum markers and the possible correlations of the between the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS (criteria 2003)
* Healthy controls

Exclusion Criteria:

* any condition mimicking PCOS
* any systematic disease

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Outpatient women with PCOS (normalweight, overweight plus obese) Healthy volunteers controls (normalweight, overweight plus obese)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
high sensitivity C-Reactive Protein (hsC-RP) levels and differences between the phenotypes | 1 hour
Lipoprotein-associated phospholipase2 (Lp-PLA2) levels and differences between the phenotypes | 1 hour
Cardiovascular Risk Assessment and differences between the phenotypes | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Second Department of Obstetrics and Gynecology, Third Department of Cardiology, Second Propedeutic Department of Internal Medicine, Aristotle University, Thessaloniki, Greece

REFERENCES:
- [Derived] Daskalopoulos G, Karkanaki A, Piouka A, Prapas N, Panidis D, Gkeleris P, Athyros VG. Excess Metabolic and Cardiovascular Risk is not Manifested in all Phenotypes of Polycystic Ovary Syndrome: Implications for Diagnosis and Treatment. Curr Vasc Pharmacol. 2015;13(6):788-800. doi: 10.2174/1567201812666150120163025. PMID 25600030